CLINICAL TRIAL: NCT03226197
Title: Feasibility and Safety of Delivering a Ketone Drink to Comatose Survivors of Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 011774
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Ketone ester drink to be administered by nasogastric tube. Initial bolus dose of 25 ml on enrollment. After 1 hour, begin 47 hr infusion at 6 ml per hour.
  Interventions: Dietary Supplement: Ketone ester drink

INTERVENTIONS:
Dietary Supplement: Ketone ester drink — Ketone ester drink

SUMMARY:
Every year, efforts are made to resuscitate about 30,000 people when their hearts stop outside of the hospital environment ('out-of-hospital cardiac arrest'). Early damage to the brain due to 'oxygen starvation' (seemingly paradoxically) gets worse when blood flow is restored. Of the 6,350 survivors admitted to intensive care units, 46% die from brain damage, and half of those who survive suffer long-term brain damage. Apart from avoiding a high temperature, nothing has been found which can protect the brain or improve outcome.

'Ketones' are chemicals naturally produced in the body from fat during starvation. They act as an energy source, but also as regulators of metabolism, and appear to protect cells from damage when oxygen supplies are scarce, or when blood flow is restored. The investigators want to see whether a ketone drink will protect the brain after out-of-hospital cardiac arrest.

The investigators will study 10 cardiac arrest patients, and participants will be given the ketone drink via a feeding tube (which is routinely passed into the stomach in such cases). The investigators shall check that the drink is absorbed, and measure the ketone levels in the blood. The investigators will also measure important aspects of blood chemistry (including pH and blood sugar) and collect data on brain (electrical recordings called 'EEG' and 'SSEP') and heart function (ultrasound scans or 'echocardiographs') - both of which it is hoped might improve - in order to demonstrate that this is possible if it is to be included in a subsequent large trial. The study will be scrutinised by world experts in the field, who have also helped design the study.

If this pilot study is a success, the investigators will apply to a major grant body to fund an appropriately-powered randomised controlled trial to determine whether ketones improve neurological outcome and survival in these patients. Results will also allow similar studies to be planned in heart attack, stroke and traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Male or female
* Comatose survivors of out-of-hospital cardiac arrest, defined as return of spontaneous circulation for at least 5 minutes with a score of <8 on the Glasgow Coma Scale
* For admission to intensive care unit for full, active treatment

Exclusion Criteria:

* Primary neurological or intracranial cause of cardiac arrest
* In-hospital cardiac arrest
* Inclusion in another trial at time of recruitment
* Over 4 hours from time of return of spontaneous circulation to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline arterial blood gas values for pH | 48 hours
Change from baseline arterial blood gas value for bicarbonate (mmol/L), | 48 hours
Change from baseline arterial blood gas value for base excess (mEq/L), | 48 hours
Change from baseline arterial blood gas value for glucose (mmol/L) | 48 hours
Change from baseline arterial blood gas value for lactate (mmol/L) | 48 hours
Change from baseline biochemistry laboratory results (full biochemistry panel including lipids, non-esterified fatty acids and serum insulin as per study protocol) | 48 hours
Change from baseline haematology laboratory results (full blood count and coagulation profile as per study protocol) | 48 hours
Time from arrival of participant to ketone drink administration (hh:mm) | 24 hours
Number of participants receiving full course of ketone drink | 48 hours
  As defined in study protocol: 25ml bolus followed after 1 hour by 47 hour infusion at 6 ml per hour
Change from baseline serum troponin (ng/ml) | 12 hours
Change from baseline serum neuron specific enolase (ng/ml) | 48 hours

SECONDARY OUTCOMES:
Change from baseline level of plasma betahydroxybutyrate (mmol/L) | 48 hours
Number of participants undergoing electroencephalogram as per protocol | 72 hours
Number of participants undergoing somatosensory evokes potentials as per protocol | 72 hours
Number of participants undergoing echocardiography as per protocol | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Jain, MBBS MD, Principal Investigator — Consultant Cardiologist
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No